CLINICAL TRIAL: NCT04039399
Title: Ischemic Conditioning Chronic Stroke Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Matthew J. Durand, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00033275
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study PI will be blinded to the intervention until after all plasma samples have been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Conditioning (Experimental): Study participants will receive one session of ischemic conditioning on their affected leg with cuff inflation to 225 mmHg.
  Interventions: Procedure: Ischemic Conditioning
- Sham Ischemic Conditioning (Sham Comparator): Study participants will receive one session of sham ischemic conditioning on their affected leg with cuff inflation to 10 mmHg.
  Interventions: Procedure: Sham Ischemic Conditioning

INTERVENTIONS:
Procedure: Ischemic Conditioning — Ischemic conditioning is a well-defined, non-invasive procedure which consists of inflating a blood pressure cuff around a limb (in our study, the paretic leg), inflating the cuff to 225 mmHg to occlude blood flow to the limb for 5 minutes, releasing the cuff for 5 minutes, and repeating 5 times. In our study, participants will receive one session of the intervention (45 minutes total).
  Arms: Ischemic Conditioning
Procedure: Sham Ischemic Conditioning — There will also be an IC Sham group which is identical to the IC intervention, except the cuff is only inflated to 10 mmHg, which is a high enough pressure to perceive cuff tightness but not high enough to have any physiological effects.
  Arms: Sham Ischemic Conditioning

SUMMARY:
Stroke is the leading cause of disability in adults in the United States. Despite advances in hyperacute stroke care, advancements in stroke rehabilitation are lagging. We have previously shown that a non-invasive, cost-effective, easy to perform intervention, called ischemic conditioning (IC), can improve paretic leg strength, reduce muscle fatigue, and increase walking speed in chronic stroke survivors (>1 year post-stroke). The IC procedure makes the paretic leg transiently ischemic (5 minutes) using a cuff inflated to 225 mmHg, and repeats the occlusion 5 times with 5 minute periods of rest between cycles (45 total minutes). It is well accepted that the response to IC is complex and involves local, humoral and neural factors. The mechanism by which IC can confer motor benefit in stroke survivors is unknown. The aim of this study is to examine if IC can increase sympathetic nervous system (SNS) activity, which would promote an increased cardiovascular response to exercise and increased muscle strength. We hypothesize that plasma epinephrine and norepinephrine levels will increase more during a cold pressor test (a well-tolerated test to induce a sympathetic response) in chronic stroke survivors who undergo a single session of IC vs. IC-Sham. To accomplish the goals of this study, 15 chronic stroke survivors will each make two visits to the adult translational research unit at Medical College of Wisconsin (MCW) to have either IC or IC-Sham performed on their paretic leg in a counterbalanced order. Venous blood will be drawn before and after the IC or IC-Sham procedure and after a two-minute cold pressor test where the study participants submerge their hand into a bucket of ice water. This will cause an increased sympathetic response, which will be assessed by measuring blood pressure and the relative increase in the levels of circulating catecholamines (epinephrine and norepinephrine, assessed by high performance liquid chromatography).

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be between 18-85 years of age, able to give informed consent, >1 year post diagnosis of unilateral cortical or sub-cortical stroke, have residual lower limb paresis.

Exclusion Criteria:

* History of blood clots in the extremities or any condition in which compression of the thigh or transient ischemia is contraindicated (e.g. wounds in the leg), chronic pain syndrome, history of head trauma, comorbid neurological disorder, any uncontrolled hypertension (>160/100 mmHg), peripheral vascular disease, a myocardial infarction in the previous year, inability to follow 2 step commands, or history of multiple strokes.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Norepinephrine Concentration | Through study completion, an average of 1 year
  We will compare the absolute change in plasma norepinephrine from immediately after IC or IC Sham to immediately after the cold pressor test (i.e. the change in concentration from rest to immediately after the cold pressor test; comparison is deltaIC vs. deltaIC Sham).

SECONDARY OUTCOMES:
Change in Plasma Epinephrine Concentration | Through study completion, an average of 1 year
  We will compare the absolute change in plasma epinephrine from immediately after IC or IC Sham to immediately after the cold pressor test (i.e. the change in concentration from rest to immediately after the cold pressor test; comparison is deltaIC vs. deltaIC Sham).
Change in Systolic Blood Pressure | Through study completion, an average of 1 year
  We will compare the absolute change in systolic blood pressure from immediately after IC or IC Sham to immediately after the cold pressor test (i.e. the change in systolic blood pressure from rest to immediately after the cold pressor test; comparison is deltaIC vs. deltaIC Sham).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04039399/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04039399/SAP_001.pdf
  • Informed Consent Form (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT04039399/ICF_002.pdf